CLINICAL TRIAL: NCT05140421
Title: Strengthening the Safety Net: Testing a Novel Data-to-Suppression (D2S) Intervention Strategy in the Ryan White HIV/AIDS Program
Brief Title: Testing a Novel Data-to-Suppression (D2S) Intervention Strategy in the Ryan White HIV/AIDS Program
Acronym: D2S
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City University of New York (Other)
Collaborators: New York City Department of Health and Mental Hygiene (Other Government); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mary Irvine, Director of HIV Care and Treatment Research and Evaluation, New York City Department of Health and Mental Hygiene
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00000707; R01MH125735 (NIH)
Record Dates: First submitted 2021-11-19; First posted 2021-12-01 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Hiv
Keywords: viral load suppression; surveillance; HIV treatment engagement; structural intervention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — dextrin 2-sulfate

STUDY DESIGN:
Intervention Model Description: Stepped-wedge design: To isolate the effects of D2S on viral suppression, the investigators will randomize (within matched pairs and one trio) 27 RWPA-funded behavioral health and housing services provider agencies to immediate or delayed implementation of D2S (12 months apart).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Implementation (Experimental): This arm will receive D2S intervention components during Period 1 (Early Implementation) as well as throughout Period 2 of the stepped-wedge trial.
  Interventions: Behavioral: Data to Suppression (D2S)
- Delayed Implementation (Active Comparator): This arm will receive no D2S intervention components during Period 1 (Early Implementation), but will then receive all D2S intervention components in Period 2, starting 12 months later.
  Interventions: Behavioral: Data to Suppression (D2S)

INTERVENTIONS:
Behavioral: Data to Suppression (D2S) — Intervention components include (1) reporting and (2) capacity building to facilitate identification of and follow-up with PWH who are in care but virally unsuppressed. The NYC Health Department will send client-level, surveillance-based reports on individual clients' viral suppression status to those clients' current Ryan White Part A behavioral health and housing service providers. The Health Department will also provide capacity building and technical assistance (TA) support to service providers on following up with clients flagged as unsuppressed, and on addressing barriers to viral suppression through root cause analyses and the development and implementation of D2S quality improvement projects. The intervention components are all delivered to Ryan White Part A providers by the Health Department, in order to enhance program resources to achieve and maintain viral suppression in the Ryan White Part A client population in NYC.

SUMMARY:
The Ryan White HIV/AIDS Program (RWHAP) for low-income people with HIV (PWH) is a key resource for reducing HIV health disparities and scaling up evidence-based interventions. As RWHAP serves >50% of US PWH, RWHAP outcomes are vital to achieving "getting-to-zero"/ Ending the HIV Epidemic (EHE) Plan targets.

As a grantee for RWHAP Part A (RWPA) funding distributed to the counties/cities severely affected by HIV, New York City (NYC) conducts regular HIV care continuum monitoring citywide and in its RWPA programs, which offer support services to reduce social and behavioral barriers to care/treatment. Local data consistently show lower viral suppression (VS) among RWPA clients in HIV care than among non-RWPA PWH in HIV care. Relative to NYC HIV cases overall, NYC RWPA clients (~14,000 per year) over-represent Black and Latinx PWH and high-poverty neighborhoods. To address local outcome disparities and to fill gaps left by data-to-care strategies and research focused on medical care (re-)linkage, the investigators propose to implement and rigorously evaluate the effectiveness of a novel 'data-to-suppression' (D2S) intervention among RWPA behavioral health and housing program clients who are in HIV care but unsuppressed. Surveillance-based reports on unsuppressed clients plus D2S capacity-building assistance will guide RWPA providers in targeting and delivering evidence-informed strategies to improve VS.

DETAILED DESCRIPTION:
The investigators will implement and evaluate the Data-to-Suppression (D2S) intervention in Aim 1, which applies a cluster-randomized, stepped-wedge design. Agencies eligible for the trial will be matched in pairs and then randomized within pairs to early (Period 1) or delayed (Period 2) D2S intervention implementation. Our design will also use baseline data from a 12-month pre-implementation period (Period 0), for which D2S reports will be retrospectively generated. Each period will include two rounds of report releases (six months apart), each with a 12-month look-back period. Period 2 will begin 12 months after the start of Period 1. In both arms, clients without viral suppression (VS) will be followed forward for viral load (VL) outcomes after report issue date. Outcomes data will be derived from the NYC HIV Surveillance Registry, a population-based data source of longitudinal laboratory (VL, CD4) testing records on all diagnosed NYC PWH, regardless of medical provider within NYC, and for periods extending before and after RWPA program enrollment or discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* For each stepped-wedge implementation period (Period 0, 1, or 2), clients eligible for trial inclusion must have: (1) ≥1 viral load (VL) test in the report year (evidence that they are in HIV care in NYC); (2) unsuppressed VL (≥200 copies/mL) at last reported VL test during that year; and (3) a reported service in one of the eligible programs/agencies during the report year. In addition, they must still have an open RWPA enrollment in one of the eligible programs and agencies and be presumed living at the time of report generation (two months following the end of the report year on which data are being shared with providers).

Exclusion Criteria:

* Agencies without current NYC RWPA funding for housing assistance or behavioral health (mental health, supportive counseling or harm reduction) services are excluded. Agencies with <5 clients meeting the above inclusion criteria over three recent pre-implementation sample periods of data are also excluded (due to insufficient numbers of unsuppressed clients). Clients enrolled in NYC RWPA behavioral health or housing programs are excluded from the trial if they are virally suppressed, deceased, or lacking any evidence of NYC HIV care for a full year at the time a D2S report is issued. Given the potential lag in reporting to surveillance and the need to use the freshest available surveillance data for D2S reports, some clients may later be found to have died or to have a VL<200 dated after their qualifying VL≥200 but prior to D2S report generation; such clients will be excluded post hoc from that round of follow-up due to VS at the time of intervention. Similarly, clients later reported (in programmatic data) to have been closed out of all eligible programs before the report issue date will be excluded post hoc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1619 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Timely viral suppression | 6 months
  Registry-reported VL <200 copies/mL on any VL test dated in the six months after the client first appeared as unsuppressed on a D2S report for the period

SECONDARY OUTCOMES:
Time to viral suppression | 12 months
  Time to first VL <200 copies/mL after client's first appearance on a D2S report for the period

CONTACTS AND LOCATIONS:
Overall Officials: Denis Nash, PhD, Principal Investigator — CUNY School of Public Health and Health Policy; Mary K Irvine, DrPH, Principal Investigator — New York City Department of Health and Mental Hygiene
Locations (27):
- United States (27):
  - Alliance for Positive Change, New York, New York
  - Mount Sinai Beth Israel, New York, New York
  - Exponents, Inc., New York, New York
  - GMHC, New York, New York
  - African Services Committee, Inc., New York, New York
  - Harlem United, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Bailey House, Inc., New York, New York
  - New York Harm Reduction Educators, Inc., New York, New York
  - The Institute for Family Health, New York, New York
  - NYC Health and Hospitals Harlem, New York, New York
  - Project Hospitality, Inc., New York, New York
  - Boom!Health, New York, New York
  - BronxWorks, Inc., New York, New York
  - St. Ann's Corner of Harm Reduction, New York, New York
  - Tolentine Zeiser Community Life Center, New York, New York
  - Housing Works, New York, New York
  - Research Foundation of State University of New York, New York, New York
  - La Nueva Esperanza, Inc., New York, New York
  - NYC Health and Hospitals Woodhull, New York, New York
  - Interfaith Medical Center, New York, New York
  - Bridging Access to Care, Inc., New York, New York
  - After Hours Project, New York, New York
  - Planned Parenthood of Greater New York, New York, New York
  - CAMBA, Inc., New York, New York
  - AIDS Center of Queens County, Inc., New York, New York
  - NYC Health and Hospitals Queens, New York, New York

IPD SHARING:
Plan to Share IPD: No
Due to New York State Public Health Law and the confidential nature of HIV surveillance data in New York, public health authorities in New York City cannot release individual-level data on reported HIV cases for purposes other than ensuring appropriate HIV care. The NYC Department of Health and Mental Hygiene (DOHMH) staff are available to assist external researchers who may have further specific data questions or uses. Please send an email to the DOHMH PI Mary Irvine (mirvine@health.nyc.gov) with questions or requests for additional information.

REFERENCES:
- [Derived] Irvine MK, Abdelqader F, Levin B, Thomas J, Avoundjian T, Peterson M, Zimba R, Braunstein SL, Robertson MM, Nash D. Study protocol for data to suppression (D2S): a cluster-randomised, stepped-wedge effectiveness trial of a reporting and capacity-building intervention to improve HIV viral suppression in housing and behavioural health programmes in New York City. BMJ Open. 2023 Jul 14;13(7):e076716. doi: 10.1136/bmjopen-2023-076716. PMID 37451738